CLINICAL TRIAL: NCT00731484
Title: Validation of TearLab Osmometer - Human Factor Usability Report
Status: Completed | Type: Observational
Sponsor: TearLab Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP00004
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Disease; Tear Osmolarity; Tear Osmolality
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteer Patients/Subjects: These subjects should present the general population.

SUMMARY:
The objective of this study is to validate the performance of the OcuSense TearLab™ osmolarity test when performed in physician office laboratories (POL) by health care professionals using human tear fluid collected from volunteer subjects and contrived tear samples.

DETAILED DESCRIPTION:
To validate the performance and usability of the TearLab osmometer, specifically human factor usability, when used in the hands of intended users, i.e. ophthalmology and optometry clinics. This testing is required to insure that the Osmolarity System meets the Product Requirements and for completion of the Technical File, Design History File and FDA 510(k) Submission.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers representing the general population (a minimum of 120 subjects representing 50% of the total study population,
* Otherwise healthy volunteers previously-diagnosed with moderate or severe chronic dry eye and/or Sjogrens syndrome and/or designated as dry eye disease subjects by the OSDI questionnaire (a minimum of 40 subjects representing 50% of the total study population),
* Men or women,
* Adult 18 years or older,
* Contact lens wearers may participate,
* Patients having undergone refractive surgery may participate,
* Patients having undergone cataract surgery may participate

Exclusion Criteria:

* Eye pathology other than previously-diagnosed moderate or severe chronic dry eye and/or Sjogrens syndrome, Use of topical medication within the last 24 hours,
* Eye drop usage within the last 2 hours,
* Ocular surface staining within the last 2 hours,
* Other invasive ocular diagnostic testing within the last 2 hours,
* Crying within the last 30 minutes,
* Eye makeup present on the eye lid within 10 minutes of tear collection,
* Examination by slit lamp within 10 minutes of tear collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmic and optometric clinics.
Sampling Method: Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lemp, MD, Study Chair — Clinical Professor of Ophthalmology, Georgetown University
Locations (3):
- United States (3):
  - Gordon Binder Weiss Vision Institute, San Diego, California
  - Kentucky Lion Eye Center, University of Louisville, Louisville, Kentucky
  - The Ohio State University College of Optometry, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The data was used in the FDA 510(K) submission.

RESULTS

PARTICIPANT FLOW:
Groups:
- General Population: Healthy normal volunteers as well as subjects diagnosed with moderate or severe chronic dry eye disease and/or Sjögrens syndrome. Subjects were recruited from among patients presenting for a routine visit at the physician office study sites.
Period: Overall Study
Arm/Group | General Population
Started | 233
Completed | 233
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | General Population
Number analyzed (Participants) | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 191
  >=65 years | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 74
Region of Enrollment [Number; unit: participants]
  United States | 233

OUTCOME MEASURES:

1. Primary Outcome: Tear Osmolarity in Human Measured by TearLab System
Description: Tear osmolarity was measured with a laboratory-on-a-chip, which simultaneously collects and analyzes the electrical impedance of a 50 nL tear sample from the inferior lateral meniscus (TearLab Osmolarity System). The results are reported in mOsm/L. The trial was not set up to evaluate diagnostic performance, as no gold-standard method was used to establish dry eye status, but rather, to determine whether the TearLab could measure tear osmolarity in human subjects.
Time Frame: Single visit, at time of tear osmolarity testing.
Population: Healthy normal volunteers as well as subjects diagnosed with moderate or severe chronic dry eye disease and/or Sjögrens Syndrome
Measure: Mean (Full Range); unit: mOsms/L
Groups:
- General Population: Subjects were recruited from patients presenting for a routine visit at the physician office study sites
Arm/Group | General Population
Number analyzed (Participants) | 233
mOsms/L | 308 [275 to 369]

ADVERSE EVENTS:
Time Frame: Time of single visit
Description: No side effects were observed or reported.
Arm/Group | General Population
Serious Adverse Events (participants affected / at risk) | 0/233
Other Adverse Events (participants affected / at risk) | 0/233

LIMITATIONS AND CAVEATS:
As recruitment came from the general clinical population, only 19 subjects were classified as having Sjögren's Syndrome, and few of the subjects had severe dry eye. Therefore, the upper range is lower than we have observed in the following studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No